CLINICAL TRIAL: NCT06410339
Title: Ultrasound Assessment of Anatomical Changes in the Fingers of Recreational Rock Climbers
Status: Recruiting | Type: Observational
Sponsor: Rocky Vista University, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-195
Record Dates: First submitted 2024-04-30; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Flexor Tendons Injuries
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- rock climbers: rock climbers of varying experience levels 18-40 years old
  Interventions: Diagnostic Test: Ultrasound
- control: non rock climbers 18-40 years old
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — ultrasound of flexor tendons on hands

SUMMARY:
The objective of this study is to assess whether recreational rock climbers experience thickening of the flexor digitorum tendon in the 2nd 3rd and 4th fingers. In these fingers the study will also assess whether there is thickening of the A2 annular pulley and if there is a measurable increase in the tendon to bone distance at the level of the A2 pulley when the fingers are placed into flexion against mild resistance. This study aims to provide clinicians with an understanding of how exposure to rock climbing can lead to chronic anatomical changes to the soft tissue structures of the finger. These changes have been demonstrated in the elite rock climber population, but have yet to be studied in the much larger and growing recreational rock climbing population which consisted of nearly 10 million participants in 2021. If significant, these anatomical variations might guide the assessment of imaging and clinical decision making when managing finger injuries in patients with exposure to rock climbing. Portable ultrasound probes will be used to scan and measure the dimensions of various soft tissue structures in the hands of both rock climbers and a control population, this data will be paired with data collected in a brief survey asking about exposure to rock climbing, history of finger injuries, and style of climbing.

DETAILED DESCRIPTION:
The aim of this study is to assess whether there in an increase in the diameter of the flexor digitorum tendon, an increase in thickness of the A2 annular pulley, and the tendon to bone distance at the A2 pulley in recreational rock climbers when compared to the general population when assessed using sonography. Recreational rock climbing is an emerging sport with more than 10 million estimated participants in the United States alone. Point of care ultrasound is a common, affordable modality to assess finger injuries and is being used commonly by sports medicine physicians globally. Measuring the ligamentous tendinous structures in the fingers is one technique used to assess inflammation or degeneration of these structures. It has been demonstrated that there are significant anatomical differences present in a population of elite-level rock climbers, but this has not yet been assessed in the much larger recreational climbing population. If this study can demonstrate that recreational rock climbers display similar anatomical changes, sports medicine physicians might consider whether or not their patient has significant exposure to this activity when assessing these structures. This study will use high frequency ultrasound (12MHz) to assess anatomic landmarks in the fingers of study participants. All data will be de identified. Statistical analysis will involve a variety of modalities including T-test, Chi square analysis and ANOVA. The data collected will be de-identified using a participant number and stored separately from all identifying data. Data will be stored in a password protected OneDrive file. Participant information will be stored in a separate password protected OneDrive file. All researchers will have access to the data collected for data analysis. Dr. Vidlock alone will have access to the participant identifying data. Data with subject identifiers will not be released to other individuals or agencies. Data collection for the experimental group in this study will be conducted at the Ubergrippen Indoor Climbing Crag in Denver, CO. Data collection for the control group in the study will be conducted at the RVU Colorado campus. Ultrasound images taken of the flexor digitorum tendon in the 2nd, 3rd, and 4th fingers will be measured onsite immediately after data collection is completed. The study will be completed in a single sitting taking approximately 10 minutes to capture ultrasound images of the 3 digits on each hand. Participants will then complete a survey that should take no longer than 10 minutes to complete. Participants will be invited to voluntary participate until approximately 25 climbers, and 25 control subjects have been assessed. Participants must be between 18-40 years old. All participants must participate in some form of exercise 2-5x per week on average. Participants will be excluded if they have been diagnosed with a ligamentous or tendinous injury in the fingers being tested. Participants will be excluded if they have a diagnosed connective tissue disorder, or any other condition affecting the structure or function of their fingers. Patients who are known to be pregnant will be excluded. Participants must be between 18-40 years old. All participants must participate in some form of exercise 2-5x per week on average. Participants will be excluded if they have been diagnosed with a ligamentous or tendinous injury in the fingers being tested. Participants will be excluded if they have a diagnosed connective tissue disorder, or any other condition affecting the structure or function of their fingers. Patients who are known to be pregnant will be excluded.

The climber group subjects must have at least 6 contiguous months of climbing experience and climb more than 2x but less than 4x per week.

The control group must have no consistent climbing experience. (less than 3x in the past 6 months, less than 10x total)

ELIGIBILITY:
Inclusion Criteria:

*Able to hold finger still for ultrasound measurement

Exclusion Criteria:

* Previous ligamentous or tendinous injury in the fingers being tested
* Connective tissue disorder
* Condition affecting the structure or function of their fingers.
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy 18-40 year olds
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Injuries to finger, specifically flexor tendon | 1 year
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Rocky Vista University, Parker, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided
Available upon request at this time

REFERENCES:
- [Background] Klauser A, Bodner G, Frauscher F, Gabl M, Zur Nedden D. Finger injuries in extreme rock climbers. Assessment of high-resolution ultrasonography. Am J Sports Med. 1999 Nov-Dec;27(6):733-7. doi: 10.1177/03635465990270060801. PMID 10569358
- [Background] El-Sheikh Y, Wong I, Farrokhyar F, Thoma A. Diagnosis of finger flexor pulley injury in rock climbers: A systematic review. Can J Plast Surg. 2006 Winter;14(4):227-31. doi: 10.1177/229255030601400405. PMID 19554140
- [Background] Schoffl V, Simon M, Lutter C. [Finger and shoulder injuries in rock climbing]. Orthopade. 2019 Dec;48(12):1005-1012. doi: 10.1007/s00132-019-03825-3. German. PMID 31705177